CLINICAL TRIAL: NCT00528684
Title: A Phase I/II Clinical Trial to Evaluate Dose Limiting Toxicity and Efficacy of Intralesional Administration of REOLYSIN® for the Treatment of Patients With Histologically Confirmed Recurrent Malignant Gliomas
Brief Title: Safety and Efficacy Study of REOLYSIN® in the Treatment of Recurrent Malignant Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oncolytics Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REO 007
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2011-09

CONDITIONS: Malignant Glioma
Keywords: Oncolytics Biotech; cancer alternative therapies; malignant glioma; glioblastoma multiforme; oncolytic virus; reovirus; REOLYSIN
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — reolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: REOLYSIN® — REOLYSIN® is administered as a single intratumoral infusion over 72 hours. Dose levels in Phase 1 will be 1x10E8, 3x10E8, 1x10E9, 3x10E9, 1x10E10 TCID50. The dose level for Phase 2 will be the top dose reached in Phase 1.

SUMMARY:
RATIONALE: Oncolytic viruses such as reovirus (REOLYSIN®) can specifically kill tumor cells while leaving healthy cells unharmed.

PURPOSE: This phase I/II study investigates the maximum tolerated dose (MTD), dose limiting toxicity (DLT) and anti-tumor effect of intralesional administration of REOLYSIN® therapeutic reovirus in patients with malignant glioma with evaluable disease which is progressive/recurrent despite surgery and/or radiotherapy with or without chemotherapy. (The phase I portion of the study is currently enrolling patients.)

DETAILED DESCRIPTION:
Oncolytic viruses, such as reovirus, are those viruses which specifically destroy cancer cells. Reovirus is a common virus that does not cause disease, and has been shown to be associated with only minor flu-like symptoms. REOLYSIN® is a formulation of the live, replication-competent wild-type reovirus that selectively replicates in tumor cells, while leaving healthy cells unharmed.

This phase I/II multi-center study follows a standard design utilizing therapeutic viral dosage escalation. The phase I portion of the trial will evaluate the doses of intralesional REOLYSIN titrated to a maximum tolerated dose (MTD). The objective of the phase II portion of the study is to assess tumor response. The proportion of patients surviving to six months and the safety of REOLYSIN® are secondary objectives.

Each patient enrolled in the study will receive a single infusion of REOLYSIN® over 72 hours. Patients will remain in hospital for at least 90 hours after initiation of infusion. Following REOLYSIN® administration, each patient will be followed for at least 12 weeks (Phase I) and at least 6 months (Phase II) with regular evaluation visits (weekly and then monthly). Evaluations will include tumor measurements, serial neurologic exams and functional performance status assessments at baseline, prior to hospital discharge, and at weeks 4, 8, 12, 16 and 24 after REOLYSIN® therapy. Changes in performance will be assessed using the Karnofsky Performance Status scale. Subjects will also undergo serial blood sampling for evaluation of viral RNA, hematology and biochemistry.

ELIGIBILITY:
Abbreviated Inclusion Criteria:

* PHASE I: 1st, 2nd or 3rd recurrence of: glioblastoma multiforme; gliosarcoma; anaplastic astrocytoma; anaplastic mixed glioma; or anaplastic oligodendroglioma
* PHASE II: 1st recurrence of glioblastoma multiforme (only)
* Progressing/recurrent lesion which is ≥1cmx1cm. For the Phase II study the lesion must be ≤5cmx5cm, defined by MRI only
* Be fully recovered from any prior therapy
* Have been treated at the time of original diagnosis by surgery and external beam radiation to a dose of at least 5000 cGy; radiotherapy completed at least 6 weeks before REOLYSIN® therapy
* Any intracranial surgery, except for stereotactic needle biopsy, must have occurred at least 4 weeks before REOLYSIN® therapy
* Any anti-cancer drug therapy must have been completed at least 4 weeks (6 weeks in the case of prior nitrosourea therapy) before REOLYSIN® therapy
* Have a life expectancy of ≥8 weeks and a Karnofsky Performance Status (KPS) of ≥60
* Absolute neutrophils ≥1.5 x10^9/L; hemoglobin ≥100g/L; platelets ≥100 x 10^9/L
* ALT ≥1.5 x ULN; total bilirubin ≥1.5 x ULN
* Serum creatinine ≤1.5 x ULN
* EKG with no evidence of active, acute cardiovascular disease
* PT within normal limit
* Women of childbearing potential must have a negative pregnancy test
* Reside or have suitable living arrangements within a reasonable geographical area of the study site and be able to participate in all follow-up visits
* Patients requiring corticosteroids must be on a stable dose of steroid for at least two weeks prior to baseline MRI and when entered in the study. Maximum daily dose of 24 mg/day of dexamethasone/decadron or equivalent

Abbreviated Exclusion Criteria:

* Patients who are sexually active and not willing to use barrier methods of contraception; women who are breastfeeding
* Patients with unstable or serious concurrent medical or psychiatric conditions that would interfere with study treatment or follow-up
* Patients with more than one discrete enhancing lesion on MRI, or radiographic evidence of satellite lesions or leptomeningeal disease not obviously contiguous by FLAIR imaging
* Patients who may require further neurosurgery within 4 weeks after REOLYSIN® treatment
* Patients with a prior history of encephalitis, multiple sclerosis or other significant chronic CNS disease
* Patients who have evidence of a current CNS infection, meningeal gliomatosis or gliomatosis cerebri
* Patients with tumor that to be treated would require needle or catheter passage through a ventricle, the posterior fossa or basal ganglia; or patients with tumors invading the ventricle
* Patients who have previously participated in experimental viral therapy protocols
* Patients who have had prior intratumoral gene therapy or other intratumoral therapies
* Patients who have had Gliadel wafer therapy less than 6 months prior to enrollment
* Patients who have a history of bleeding disorders including congenital or acquired coagulopathies
* Patients who have a known history of hepatitis or tuberculosis
* Patients who have a known history of hereditary or acquired immunodeficiency including HIV infection
* Patients who have impaired non-neurological organ function (>Grade 1)
* Patients who have used systemic antiviral (or potentially antiviral) therapies within 28 days of enrollment
* Patients who have had brachytherapy or radiosurgery to the brain at any time
* Patients with previous or concurrent malignancies at other sites (except surgically-cured carcinoma in situ of the cervix and non-melanoma skin cancer)
* Prior or current medical history indicating that a patient may be significantly immunosuppressed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-07; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
determine the maximum tolerated dose | in the first 28 days following REOLYSIN® administration
and response rate of treated tumors | evaluated monthly for 6 months following REOLYSIN® administration
determine the dose limiting toxicity | in the first 28 days following REOLYSIN® administration

SECONDARY OUTCOMES:
Determine the patient survival | patients are in follow up for up to six months
functional status using the Karnofsky Performance Status scale and Clinical Neurological Assessment | evaluated monthly for up to 6 months
time to progression for the treated tumor | evaluated monthly for up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: James M Markert, MD, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - The Ohio State University Medical Center and Arthur G. James Cancer Hospital and Richard J. Solove Research Center, Columbus, Ohio